CLINICAL TRIAL: NCT05477745
Title: The Correlation Between Femoral Component Implanting Flexion Angle and Posterior Condyle Offset in Cruciate Retaining Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2022-0048
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Knee Osteoarthritis
Keywords: Sagittal flexion angle; Posterior femoral offset; Cruciate-retaining total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The group that the sagittal flexion angle of the femoral component less than 4°: The patients' knees were taken on the X-ray examination after the total knee arthroplasty on the medial-lateral position. The flexion (positive degree) or extension (negative degree) angle of the femoral component according to the anterior femoral cortex was measured. The patients with the sagittal flexion angle of the femoral component less than 4° were categorized into this group.
  Interventions: Procedure: total knee arthroplasty
- The group that the sagittal flexion angle of the femoral component over 4°: The patients' knees were taken on the X-ray examination after the total knee arthroplasty on the medial-lateral position. The flexion (positive degree) or extension (negative degree) angle of the femoral component according to the anterior femoral cortex was measured. The patients with the sagittal flexion angle of the femoral component over 4° were categorized into this group.
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total knee arthroplasty — The surgeries were performed under general anesthesia. The medial parepatellar incision was introduced during the TKA. The femoral component size was selected according to the intro-operative measurement. The osteotomy was done according to the intramedullary guide and the cutting guide. After the proximal tibial osteotomy was finished, the cruciate-retaining Total Knee System was used. The lateral rotation of the femoral component was determined by the gap-balancing technique.

SUMMARY:
The main aim and scope is making measurement and comparison about the femoral component posterior offset under different femoral component implanting flexion angle in cruciate retaining total knee arthroplasty. The results may identify the influence of the flexion component implanting flexion angle on the femoral component posterior offset.

ELIGIBILITY:
Inclusion Criteria:

* The patients undertaken the primary cruciate retaining total knee arthroplasty;
* using the curiate retaining total knee arthroplasty prothesis from Biomet and Smith&Nephew;
* Complete surgery documents and radiologic data,such as standard X-ray postoperative both at antirior-posterior position and medial-lateral position(overlap of the medial and lateral femoral condyle).

Exclusion Criteria:

* The patients without standard X-ray postoperative both at antirior-posterior position and medial-lateral position(poor overlap of the medial and lateral femoral condyle);
* Complex primary total knee arthroplasty, using extra component such as trabecular metal,stem or et al.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients were treated with primary total knee arthroplasty in Renji Hospital affiliated to Shanghai Jiaotong University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-29 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-08-22 (Estimated)

PRIMARY OUTCOMES:
Posterior Femoral Offset | 1 week after the surgery
  The posterior femoral offset was defined as the maximal thickness of the posterior condyle projecting posteriorly to a straight line drawn as the extension of the posterior femoral shaft cortex on the medial-lateral position of the X-ray examination.
Posterior Femoral Offset Ratio | 1 week after the surgery
  The posterior femoral offset ratio was defined as the maximal thickness of the posterior condyle projecting posteriorly to a straight line drawn as the extension of the posterior femoral shaft cortex, divided by the maximal thickness of the posterior condyle projecting posterior to a straight line drawn as the extension of the anterior femoral shaft contex on the medial-lateral position of the X-ray examination.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No